CLINICAL TRIAL: NCT04142034
Title: Feasibility Trial of the iAMHealthy Intervention for Healthy Weight in Rural Children Recruited From Primary Care Clinics
Brief Title: Feasibility Trial of the iAMHealthy Intervention
Acronym: iAmHealthy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IDeA States Pediatric Clinical Trials Network (Network)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 249932; U24OD024957 (NIH)
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Results first posted 2022-08-22 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Rurality
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This feasibility trial is a multisite, RCT with two parts. In part 1, sites will be randomized into the order in which two recruitment methods, traditional or consecutive, are used to recruit study participants. In part 2, recruited participants will be randomized to receive a newsletter or newsletter plus the iAmHealthy behavioral intervention.
Who Masked: Investigator
Masking Description: Each clinics will recruit up to 28 child/caregiver pairs.The site awardee investigators will be blinded. The site awardee investigator will also identify a back-up,research-trained blinded assessor from the awardee site. The blinded coordinator will not have access to clinic charts. The clinic coordinator will instruct participants not discuss the trial or previous weights/data collected. He or she, or the designated backup, will take the height and weight measurements at baseline and six months. In case the ISPCTN site-awardee coordinator is accidentally unblinded, the backup assessor will take over all assessments for that participant.
  At each measurement time point, the blinded assessor will enter data into the electronic data capture system only for that time point-the system will blind them to data from any/all other data-collection time points. The blinded site coordinator will perform the 24-hour food recalls at recruitment and six months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- iAmHealthy Behavioral Intervention (Experimental): This intervention will receive the American Academy of Pediatrics (AAP) newsletter, group and individual sessions with the iAmHealthy behavioral intervention team via an electronic tablet provided by the sponsor.
  Interventions: Behavioral: the iAmHealthy Behavioral Intervention
- NewsLetter intervention (Active Comparator): This intervention arm will only receive the American Academy of Pediatrics (AAP) newsletter for six months.
  Interventions: Behavioral: Newsletter only arm
- Consecutive Recruitment method (Other): Using this recruitment method, clinics will identify potential eligible study participants through their medical records among those that have been seen in the clinic within the past year and those children with upcoming appointments and approach them and their caregivers about enrolling in the study.
  Interventions: Other: Consecutive Recruitment
- Traditional Recruitment method (Other): Flyers, advertisements, and other materials will be used to recruit potential participants to the study.
  Interventions: Other: Traditional Recruitment

INTERVENTIONS:
Behavioral: the iAmHealthy Behavioral Intervention — iAmHealthy Behavioral Intervention Arm
  Child/caregiver pairs in the iAmHealthy behavioral intervention arm will receive:
  * usual care at their clinic for all issues, including overweight and obesity;
  * a monthly newsletter that focuses on general child health. The child/caregiver pairs will receive six newsletters (one per month) during the six month intervention period (same newsletter provided to the newsletter-only intervention participants);
  * weekly group sessions for the first three months, followed by monthly group sessions during the next three months, for a total of 15 group sessions. The trial's iAmHealthy behavioral intervention psychologist or social worker (one team per clinic) will deliver these group sessions via an electronic tablet that the trial sponsor will supply;
  * 11 hours of individual "homework" sessions with the iAmHealthy behavioral intervention dietician
  Arms: iAmHealthy Behavioral Intervention
Behavioral: Newsletter only arm — Newsletter arm participants will receive a monthly newsletter on maintaining a healthy weight through diet and exercise
  Arms: NewsLetter intervention
Other: Consecutive Recruitment — Recruitment of study participants through identifying potential participants through their medical records
  Arms: Consecutive Recruitment method
Other: Traditional Recruitment — Recruitment of potential participants through flyers and advertisements
  Arms: Traditional Recruitment method

SUMMARY:
This research study is being done to find out which of 2 ways works best to get rural participants interested in joining a research study about children who weigh more than is considered healthy. One method researchers will use is the traditional method of reaching out to potential participants. The traditional method includes using flyers, posters, and booklets. The other method will be to target people who might be especially interested in the study. The second method uses medical records to find potential participants who are most likely to qualify for the study. This study is also being done to what works to help keep participants in a study like this.

Another goal of the study is to find out what methods work well to help get and keep children's and caregiver's weight in the healthy range. Researchers also want to see what works well to help children with a high Body Mass Index be more physically active and to eat healthier foods. The test methods researchers will use for this part of the study are (1) newsletters only and (2) newsletters plus online meetings. Participants will be randomly assigned to 1 of the 2 groups (newsletter or newsletter plus meetings.)

The newsletter-only group will receive monthly newsletters about children's health; this group will receive these letters for 6 months. The 'newsletter plus meeting group' will also receive the same monthly newsletter for 6 months. The latter group will also have online meetings with other children and adults as well as a group leader. Those in the 'newsletter plus meeting group' will also individually meet with a dietician.

This study will involve children and one of their caregivers (parent/guardian). The child and caregiver must live in a rural area. The child must be 6 to 11 years old. The child must be considered to have an unhealthy weight (high Body Mass Index). Both the child and caregiver must speak English. Up to 224 children will enter into this study. Participants will be consented through 4 different sites that are part of the IDeA States Pediatric Network.

DETAILED DESCRIPTION:
Conduct a multisite feasibility trial for the iAmHealthy intervention with two randomized controlled recruitment options (consecutive recruitment and traditional recruitment). We will examine retention, dose, and blinding that will inform the development of a larger, treatment-outcome fully powered randomized controlled trial (RCT) of the iAmHealthy behavioral intervention in the IDeA States Pediatric Clinical Trials Network (ISPCTN).

The study team will perform the iAmHealthy trial will be performed in four ISPCTN site-awardee states. Specifically, the study team will perform the iAmHealthy trial in one clinic per state.

Randomization of recruitment options occurs at the clinic level. Each clinic, in a randomly ordered sequence, will implement two methods of recruitment. Recruitment of Participants, for more detail on the two methods of recruitment.

Randomization of participants into intervention arms will occur at the individual level.

Newsletter-only Intervention Arm

Child/caregiver pairs in the newsletter-only intervention arm will receive:

* usual care at their clinic for all issues, including overweight and obesity;
* a monthly newsletter that focuses on general child health. The child/caregiver pairs will receive six newsletters (one per month) during the six month intervention period.

iAmHealthy Behavioral Intervention Arm

Child/caregiver pairs in the iAmHealthy behavioral intervention arm will receive:

* usual care at their clinic for all issues, including overweight and obesity;
* a monthly newsletter that focuses on general child health. The child/caregiver pairs will receive six newsletters (one per month) during the six month intervention period (same newsletter provided to the newsletter-only intervention participants);
* weekly group sessions for the first three months, followed by monthly group sessions during the next three months, for a total of 15 group sessions. The trial's iAmHealthy behavioral intervention psychologist or social worker (one team per clinic) will deliver these group sessions via an electronic tablet that the trial sponsor will supply;
* 11 hours of individual "homework" sessions with the iAmHealthy behavioral intervention dietician.

The iAmHealthy behavioral intervention psychologists/social worker will individualize group sessions and the iAmHealthy behavioral intervention dietician will adapt individual sessions by focusing on local cultural, religious, and ethnic factors relevant to the recommended changes in eating and activity habits. The iAmHealthy behavioral intervention includes 26 contact hours (15 hours of group sessions and 11 hours of individual sessions).

This feasibility trial will provide information toward the implementation of a fully powered, multisite, randomized behavior intervention trial that will compare the effectiveness of the iAmHealthy behavioral intervention to a newsletter-only intervention for the treatment of obesity among rural and underserved children and their primary caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. Child is rural. The child lives in a rural area, as defined by the United States Department of Agriculture (USDA) Rural Urban Commuting Area (RUCA) codes (greater than or equal to 4). We will calculate this using the 2010 Zip Code, RUCA Code crosswalk.
2. Child is ages 6-11 years at the time of consent. At the time of consent, a child must be 6 to 11 years of age. A narrow age range is necessary to decrease developmental variability. Clinics may enroll a child no earlier than her or his sixth birthday (6 years, 0 months, 0 days), and may enroll a child up to her or his 12th birthday (11 years, 11 months, 30 days).
3. Child BMI percentile is ≥85th. We will use the 85th percentile as a minimal cutoff for participation, as this is the minimal criteria for the definition of overweight. There is no upper limit on BMI percentile for inclusion.
4. Child and primary caregiver speak English. For the initial feasibility pilot, we will ask that both the child and primary caregiver speak English. For the larger trial that will follow, we will accommodate Spanish-speaking participants.
5. For the iAmHealthy behavioral intervention arm, the child and primary caregiver are available when the behavioral intervention team offers the intervention for the participating clinic. The child and primary caregiver must be available for most of the iAmHealthy behavioral intervention sessions when the behavioral intervention psychologist/social worker offers the group sessions at the participants' clinic. The behavioral team will conduct these sessions via video conference and families will attend via tablets.

   -

Exclusion Criteria:

1. Child has a physical limitation or injury that substantially limits physical mobility or has a planned medical treatment during the course of the trial that will substantially limit physical mobility. Because this trial recommends physical activity, we will exclude children who cannot comply with this health behavior.
2. Child has a known medical issue that could affect protocol compliance (e.g., cancer). If a child has a significant medical issue known to the clinic that could affect protocol compliance, we will exclude this child, as the protocol involves an intense intervention commitment.
3. Child and/or primary caregiver has a developmental delay or cognitive impairment that could affect protocol compliance. We will exclude primary caregivers and/or children with a known developmental delay, as this could negatively affect participation and measurement completion.
4. Child is enrolled in a weight-loss trial. If a child is enrolled in a weight-loss trial, we will exclude the child to avoid cross-pollination of trial interventions.
5. Child has a sibling who has already enrolled in the trial. If multiple children from the same family attempt to enroll, the statistical team will randomly select one child for enrollment. We will always allow siblings to attend the intervention, but we will not officially enroll them.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Davis, PhD, Principal Investigator — University of Kansas Medical Center; Paul Darden, MD, Principal Investigator — University of Arkansas
Locations (4):
- United States (4):
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Medical University of South Carolina, Charleston, South Carolina
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
We will conduct this trial in accordance with the following publication and data sharing policies and regulations:
  * NIH Public Access Policy. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive PubMed Central upon acceptance for publication.
  * ISPCTN Publications and Presentations Policy, which ensures accurate, responsible, and efficient communication of findings from ISPCTN clinical trials. The ISPCTN Steering Committee has approved and ratified the ISPCTN Publications and Presentations Policy, which includes representatives from all site awardees, as well as representatives from the NIH and the DCOC.
  * NIH Data Sharing Policy and the policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission Rule. Other researchers my request data from this trial by contacting Jeannette Lee, PhD, at the DCOC.
Supporting Information: Study Protocol, ICF
Time Frame: Per data and sharing polices of National Institute of Health (NIH) and the IDeA States Pediatric Clinical Trials Network (ISPCTN).
Access Criteria: To be announced (TBA)

REFERENCES:
- [Background] Davis AM, Darden PM, Snowden J, Simon AE, McCulloh RJ, Bimali M, Lee J. Rationale and protocol for a cluster randomized, cross-over trial of recruitment methods of rural children in primary care clinics: A feasibility study of a pediatric weight control trial in the IDeA States Pediatric Clinical Trials Network. Contemp Clin Trials. 2021 Aug;107:106476. doi: 10.1016/j.cct.2021.106476. Epub 2021 Jun 9. PMID 34118426
- [Derived] Zhang E, Davis AM, Jimenez EY, Lancaster B, Serrano-Gonzalez M, Chang D, Lee J, Lai JS, Pyles L, VanWagoner T, Darden P. Validation of remote anthropometric measurements in a rural randomized pediatric clinical trial in primary care settings. Sci Rep. 2024 Jan 3;14(1):411. doi: 10.1038/s41598-023-50790-1. PMID 38172325
- [Derived] Nguyen L, Phan TL, Falini L, Chang D, Cottrell L, Dawley E, Hockett CW, VanWagoner T, Darden PM, Davis AM. Rural Family Satisfaction With Telehealth Delivery of an Intervention for Pediatric Obesity and Associated Family Characteristics. Child Obes. 2024 Apr;20(3):147-154. doi: 10.1089/chi.2022.0210. Epub 2023 Apr 10. PMID 37036783
- [Derived] Darden PM 2nd, Davis AM, Lee JY, Bimali M, Simon AE, Atz AM, Lim CS, Phan TT, Roberts JR, McCulloh RJ, Pyles L, Shaffer M, Snowden JN. Active vs Traditional Methods of Recruiting Children for a Clinical Trial in Rural Primary Care Clinics: A Cluster-Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2244040. doi: 10.1001/jamanetworkopen.2022.44040. PMID 36445709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (children) were recruited through two approached: consecutive recruitment method or traditional recruitment method. The data shown for these methods is the number of individuals approached about the clinical trial and the number who were successfully recruited into the clinical trial and randomized into one of the two intervention arms
  Caregivers are not participant but are evaluated for efficacy in terms of body mass index
Groups:
- iAmHealthy + Newsletter Behavorial Intervention: This intervention will receive the American Academy of Pediatrics (AAP) newsletter, group and individual sessions with the iAmHealthy behavioral intervention team via an electronic tablet provided by the sponsor.
  the iAmHealthy Behavioral Intervention: iAmHealthy Behavioral Intervention Arm
  Child/caregiver pairs in the iAmHealthy behavioral intervention arm will receive:
  * usual care at their clinic for all issues, including overweight and obesity;
  * a monthly newsletter that focuses on general child health. The child/caregiver pairs will receive six newsletters (one per month) during the six month intervention period (same newsletter provided to the newsletter-only intervention participants);
  * weekly group sessions for the first three months, followed by monthly group sessions during the next three months, for a total of 15 group sessions. The trial's iAmHealthy behavioral intervention psychologist or social worker (one team per clinic) will deliver these group sessions via an electronic tablet that the trial sponsor will supply;
  * 11 hours of individual "homework" sessions with the iAmHealthy behavioral intervention dietician
Period: Recruitment Period
Arm/Group | Consecutive Recruitment Method | Traditional Recruitment Method | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Started | 535 | 23 | 0 | 0
Completed | 99 (The recruitment period included a hiatus in recruitment due to the pandemic) | 5 (The recruitment period included a hiatus in recruitment due to the pandemic) | 0 (the intervention arm is only relevant during period 2) | 0 (intervention arm is only relevant in period 2)
Not Completed | 436 | 18 | 0 | 0
Period: Intervention Period
Arm/Group | Consecutive Recruitment Method | Traditional Recruitment Method | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Started | 0 (Recruitment method is only relevant in period 1) | 0 (Recruitment method is only relevant in period 1) | 52 (There were 104 participants recruited into the intervention part of the study; half were randomized to the iAmHealthy + newsletter behavioral intervention.) | 52 (There were 104 participants recruited into the intervention part of the study; half were randomized to the Newsletter intervention.)
Completed | 0 | 0 | 45 | 50
Not Completed | 0 | 0 | 7 | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is participants who were recruited to the study and randomized to one of the two interventions: iAmHealthy + Newsletter behavioral intervention or newsletter intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (1.7) | 9.2 (1.7) | 9.3 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 26 | 58
  Male | 20 | 26 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 45 | 49 | 94
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 8 | 24
  White | 33 | 35 | 68
  More than one race | 3 | 8 | 11
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 52 | 52 | 104
Child body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: The participant population excludes participants from a site with data quality issues for height and weight, and participants who did not have post-intervention measurements
  kg/m^2
    number analyzed (Participants) | 34 | 39 | 73
    (all) | 26.15 (5.52) | 23.04 (3.71) | 24.48 (4.87)
Child body mass index adjusted for age and sex [Mean (Standard Deviation); unit: z-score] — Population: The participant population excludes participants from a site with data quality issues for height and weight, and participants who did not have post-intervention measurements
  z-score
    number analyzed (Participants) | 34 | 39 | 73
    (all) | 2.56 (1.41) | 1.86 (0.55) | 2.19 (1.09)
Caregiver body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: The participant population excludes participants from a site with data quality issues for height and weight, and participants who did not have post-intervention measurements
  kg/m^2
    number analyzed (Participants) | 34 | 39 | 73
    (all) | 35.54 (9.93) | 34.97 (8.48) | 35.24 (9.12)
Daily sweetened drink servings [Mean (Standard Deviation); unit: daily sweetened drink servings] — Population: Analysis population includes participants who have post-intervention measurements
  daily sweetened drink servings
    number analyzed (Participants) | 43 | 50 | 93
    (all) | 1.16 (1.30) | 1.18 (1.20) | 1.17 (1.24)
Daily fruit and vegetable servings [Mean (Standard Deviation); unit: daily fruit and vegetable servings] — Population: Analysis population is participants with post-intervention measures
  daily fruit and vegetable servings
    number analyzed (Participants) | 43 | 50 | 93
    (all) | 2.42 (1.21) | 2.62 (1.43) | 2.53 (1.33)
Daily servings of red foods [Mean (Standard Deviation); unit: daily servings of red foods] — Red foods are defined as those with greater than or equal to 7 grams of fat and/or greater than or equal to 12 grams of sugar per serving. Population: Analysis population includes participants with post-intervention measurements
  daily servings of red foods
    number analyzed (Participants) | 43 | 50 | 93
    (all) | 6.30 (1.83) | 6.39 (2.11) | 6.35 (1.97)
Average daily minutes of moderate to vigorous physical activity [Mean (Standard Deviation); unit: daily minutes of MVPA] — Daily minutes of moderate to vigorous physical activity (MVPA) information was measured using an actigraph Population: Analysis population excluded participants from a site where there were concerns regarding actigraph data quality, and participants who did not have post-intervention measures
  daily minutes of MVPA
    number analyzed (Participants) | 27 | 31 | 58
    (all) | 38.92 (36.92) | 55.46 (62.70) | 47.76 (52.54)
MVPA (%) [Mean (Standard Deviation); unit: percentage of time] — This measure is the percent of time that the participant was wearing the activity monitor that he/she was engaged in moderate to vigorous physical activity (MVPA). Population: Analysis population excludes participants from a site where there were data quality issues from the actigraph, and participants without post-intervention measurements
  percentage of time
    number analyzed (Participants) | 21 | 27 | 48
    (all) | 5.15 (2.58) | 6.13 (3.45) | 5.70 (3.11)

OUTCOME MEASURES:

1. Primary Outcome: Participant Recruitment Rate
Description: Measure participant recruitment rate for both recruitment options
Time Frame: 1 month for each recruitment option plus a 1 month catch-up period
Population: Potential study participants who were approached about the study using one of the two recruitment methods
Measure: Count of Participants; unit: Participants
Arm/Group | Consecutive Recruitment Method | Traditional Recruitment Method
Number analyzed (Participants) | 535 | 23
Participants | 99 | 5

2. Secondary Outcome: Participant Retention
Description: Calculate participant retention as the percent of randomized participants who remain in the study through the final measurement point.
Time Frame: 6 months
Population: Study participants who were randomized to one of the two behavioral interventions
Measure: Count of Participants; unit: Participants
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Number analyzed (Participants) | 52 | 52
Participants | 45 | 50

3. Secondary Outcome: Change in Child Body Mass Index From Baseline to Post-intervention
Description: This measure is derived from subtracting the child body mass index (BMI) taken at baseline from the child BMI taken at the end of the intervention period
Time Frame: 6 months
Population: Participants who had child BMI measurements at baseline and at the end of the intervention period and were at sites that did not have data quality issues with height and weight measurements.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Number analyzed (Participants) | 34 | 39
kg/m^2 | 0.32 (2.42) | 1.25 (2.22)

4. Secondary Outcome: Change in Child BMI Adjusted for Age and Sex From Baseline to Post-intervention
Description: This measure is derived from subtracting the child BMIz taken at baseline from the child BMIz adjusted for age and sex at the end of the intervention period. The BMIz is the body mass index adjusted for sex and age, and is a z-score normalized for the mean and standard deviation of the body mass index for the child's age and sex. A BMI z-score over 1.96 indicates that the child's body mass index is above the 95th percentile for his/her age.
Time Frame: 6 months
Population: Participants who had child BMI adjusted for age and sex measurements at baseline and at the end of the intervention period and were at sites that did not have data quality issues with height and weight measurements.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Number analyzed (Participants) | 34 | 39
z-score | -0.11 (0.53) | 0.12 (0.48)

5. Secondary Outcome: Change in Caregiver Body Mass Index From Baseline to Post-intervention
Description: The baseline caregiver body mass index (BMI) is subtracted from the caregiver BMI taken at the end of the intervention period
Time Frame: 6 months
Population: Participants who had caregiver BMI measurements at baseline and at the end of the intervention period and were from sites that did not have data quality issues with height and weight measurements.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Number analyzed (Participants) | 34 | 39
kg/m^2 | -0.32 (3.19) | -0.90 (3.60)

6. Secondary Outcome: Change in Daily Servings of Sweetened Drinks
Description: This measure is difference in the daily servings of sweetened drinks consumed from baseline to the end of the intervention period
Time Frame: 6 months
Population: Participants for whom data on the daily servings of sweetened drinks consumed was available at baseline and at the end of the intervention period
Measure: Mean (Standard Deviation); unit: daily servings of sweetened drinks
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Number analyzed (Participants) | 43 | 50
daily servings of sweetened drinks | 0.80 (0.72) | 0.81 (0.65)

7. Secondary Outcome: Change in Number of Servings of Fruits and Vegetables Consumed Daily From Baseline to Post-intervention
Description: This measure is the change in the number of servings of fruits and vegetables consumed daily from baseline to after the intervention period
Time Frame: 6 months
Population: Participants for whom data on the number of servings of fruits and vegetables consumed daily was available at baseline and at the end of the intervention period
Measure: Mean (Standard Deviation); unit: Daily fruit/vegetable servings
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Number analyzed (Participants) | 43 | 50
Daily fruit/vegetable servings | 0.36 (1.91) | 0 (1.78)

8. Secondary Outcome: Change in Number of Red Food Servings Consumed Daily From Baseline to Post-intervention
Description: This measure shows the change in the number of red food servings consumed daily from baseline to after the intervention period. Red foods are defined as those with greater than or equal to 7 grams of fat and/or greater than or equal to 12 grams of sugar per serving.
Time Frame: 6 months
Population: Participants for whom information on the number of daily servings of red food were available at baseline and post-intervention
Measure: Mean (Standard Deviation); unit: daily red food servings
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Number analyzed (Participants) | 43 | 50
daily red food servings | -0.78 (1.95) | -0.45 (2.56)

9. Secondary Outcome: Change in the Daily Minutes Spent in Moderate to Vigorous Physical Activity (MVPA) From Baseline to Post-intervention
Description: The number of minutes spent in moderate to vigorous physical activity (MVPA) is measured using an activity monitor worn by the participant. This measure is the change in minutes in MVPA from baseline to after the intervention period
Time Frame: 6 months
Population: Participants for whom baseline and post-intervention measurements of minutes of MVPA were available at baseline and post-intervention and were at sites without data quality issues related to activity monitors.
Measure: Mean (Standard Deviation); unit: daily minutes of MVPA
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Number analyzed (Participants) | 27 | 31
daily minutes of MVPA | -14.64 (39.88) | -28.74 (65.61)

10. Secondary Outcome: Change in the % of Time Spent in Moderate to Vigorous Physical Activity (MVPA ) While Wearing Activity Monitor From Baseline to Post-intervention
Description: The denominator for this measure is the number of minutes that the participant is wearing the activity monitor. The % of moderate to vigorous physical time (MVPA) is the percent of that time that the participant is spent in moderate to vigorous physical activity. This measure describes the change in that percent of time from baseline to after intervention.
Time Frame: 6 months
Population: Participants for whom the % of MVPA was available from the activity monitor at baseline and post-intervention and were at sites that did not have data quality issues with the activity monitors.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Number analyzed (Participants) | 21 | 27
percentage of time | -0.79 (2.71) | -1.60 (2.13)

11. Other Pre Specified Outcome: Participants in the iAmHealthy+ Newsletter Behavioral Intervention Who Receive at Least 80% of the Planned Intervention
Description: Participants who receive at least 80% of the planned intervention (dose) among those participants randomized to the iAmHealthy behavioral intervention arm who are retained through the final measurement.
Time Frame: 6 months
Population: The analysis population is the study participants randomized to the iAmHealthy + Newsletter behavioral intervention who were retained through the 6-month intervention period
Measure: Count of Participants; unit: Participants
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention
Number analyzed (Participants) | 45
Participants | 29

12. Other Pre Specified Outcome: Staff Blinding
Description: Blinding index as described by Bang (Bang et cl. Assessment of blinding in clinical trials. Control Clin Trials 2004: 25(2):143-156. It ranges from -1 to 1 where a value of 0 indicates fully successful blinding; a value of 1 indicates lack of blinding meaning that individuals were able to correctly identify participants' assigned intervention, and -1 indicates that individuals typically guessed the incorrect assignment.
Time Frame: 6 months
Population: Participants who were randomized to one of the two behavioral interventions
Measure: Mean (Standard Deviation); unit: index
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
Number analyzed (Participants) | 52 | 52
index | 0.12 (0.13) | 0.02 (0.13)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Using standard definitions of adverse events, adverse events were reported during the intervention period.
  All-cause mortality, serious and other (not including serious) adverse events were not reporting during the recruitment period for those in the consecutive recruitment or traditional recruitment arms.
Arm/Group | iAmHealthy + Newsletter Behavorial Intervention | NewsLetter Intervention
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 1/52 | 0/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iAmHealthy + Newsletter Behavorial Intervention (N=52) | NewsLetter Intervention (N=52)
Upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | NA — Broken elbow after participant increased physical activity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT04142034/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT04142034/ICF_001.pdf